CLINICAL TRIAL: NCT00889629
Title: Pilot Study: Effects of Hectorol (Doxercalciferol) Vitamin D Replacement on Proteinuria, PTH Level and Bone Turnover in Stable Kidney Transplant Recipients: a Single-Blind, Placebo-Controlled Study in Patients Receiving 25-OH Vitamin D3
Brief Title: Pilot Study Evaluating Doxercalciferol Replacement Therapy in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mariana Markell (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Mariana Markell, Prinicipal Investigator, State University of New York - Downstate Medical Center
Organization: State University of New York - Downstate Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-080
Record Dates: First submitted 2009-04-23; First posted 2009-04-29 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-01

CONDITIONS: Chronic Kidney Disease; Kidney Transplantation
Keywords: kidney transplantation; kidney transplant recipients
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — 1 alpha-hydroxyergocalciferol; 19-nor-hexafluoride vitamin D3; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxercalciferol (Experimental): Patients are randomized using an A B C D randomization scheme in which the patient and the primary investigator are blinded but the study staff is not. Active group receives doxercalciferol (Hectorol) 1mcgwith active titration based on intact PTH plus 25-OH Vitamin D3 (cholecalciferol) 400 IU. Safety labs and end point labs are monitored as per protocol, with the opportunity to increase the dose of doxercalciferol if target PTH value is not achieved by the predetermined midpoint.
  Interventions: Drug: Doxercalciferol; Drug: 25-OH Vitamin D3
- Cholecalciferol (Placebo Comparator): Patients are randomized using an A B C D randomization scheme in which the patient and the primary investigator are blinded but the study staff is not. Group 2 receives placebo (dummy bottle with pills resembling doxercalciferol) plus 25-OH Vitamin D3 (cholecalciferol) 400IU. Safety labs and end point labs are monitored as per protocol, with the opportunity to increase the dose of doxercalciferol placebo if target PTH value is not achieved by the predetermined midpoint.
  Interventions: Drug: placebo; Drug: 25-OH Vitamin D3

INTERVENTIONS:
Drug: Doxercalciferol — Active group receives doxercalciferol (Hectorol) 1mcg
  Other Names: Hectorol (the other name for Doxercalciferol)
  Arms: Doxercalciferol
Drug: placebo — Group 2 receives placebo (dummy bottle with pills resembling doxercalciferol)
  Other Names: Placebo for doxercalciferol
  Arms: Cholecalciferol
Drug: 25-OH Vitamin D3 — All groups received cholecalciferol
  Other Names: (cholecalciferol)

SUMMARY:
People with kidney transplants often develop bone disease. One reason for bone disease may be overactivity of a gland in the neck called the parathyroid gland. Overactivity of the parathyroid gland may be caused by lack of Vitamin D in the body. It has recently been discovered that many patients with kidney transplants have low Vitamin D levels. The investigators are examining the effects of doxercalciferol on parathyroid hormone levels, proteinuria and bone turnover markers in people who have had a kidney transplant.

DETAILED DESCRIPTION:
People with kidney transplants often develop bone disease. One reason for bone disease may be overactivity of a gland in the neck called the parathyroid gland. Overactivity of the parathyroid gland may be caused by lack of Vitamin D in the body. It has recently been discovered that many patients with kidney transplants have low Vitamin D levels.

25-OH Vitamin D3 is now recommended to treat kidney transplant patients with low vitamin D levels but it may not be enough to treat the parathyroid problems and bone disease. Doxercalciferol is a form of Vitamin D that has been used to treat bone disease and parathyroid problems in dialysis patients but has not yet been studied in patients with kidney transplants. We are interested in seeing whether doxercalciferol given together with 25-OH Vitamin D3 will be a better treatment for the overactive parathyroid gland and bone disease than 25-OH Vitamin D3 alone in patients with kidney transplants.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both genders between the ages of 18 and 65.
* Kidney transplant at least 1 year prior to enrollment
* Creatinine value of <2.5 mg/dl with no excursion >0.5 within the past 3 months
* Proteinuria of 500 mg/24 hours or a protein/creatinine ratio of 0.5 or greater
* Hypovitaminosis D, as defined by a 25-OH Vitamin D value of <25 ng/ml
* Intact PTH value between 150 and 600 pg/ml

Exclusion Criteria:

* History of parathyroidectomy
* History of prior intolerance to vitamin D therapy (not including hypercalcemia)
* History of biopsy proven acute rejection over the 3 months preceding enrollment
* Recent (over the past month) addition of an ACE inhibitor or Angiotensin -
* Receptor Blocking agent - patients who have been on a stable dose are acceptable
* Current use of active Vitamin D supplement (patients in whom therapy has been discontinued more than 1 month prior to enrollment are acceptable)
* Postmenopausal woman or women receiving hormone replacement therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
- iPTH value of 100 pg/ml or lower | 6 months
  The number of patients achieving the target iPTH value of 100 pg/ml or lower measured. Change in the level of iPTH (baseline as compared with 3 and 6 months) using both absolute value and percent change from baseline.

SECONDARY OUTCOMES:
Change in 1,25 D2 and D3, 25-OH Vitamin D3 levels | 6 months
  The Change in the levels of 1,25 D2 and D3, 25-OH Vitamin D3 levels (baseline as compared with 3 month and end of study)
Change in FGF-23 levels | 6 months
  The Change in FGF-23 levels (baseline as compared with 3 and 6 months) were measured.
Change in serum bone turnover markers | 6 months
  The Change in the levels of serum osteocalcin, bone alkaline phosphatase and n-telopeptide of Type I collagen levels (baseline versus 3 and 6 months
Change in Protein/creatinine ratio | 6 months
  Change in the level of Protein/creatinine ratio and or 24 hour urine for protein (baseline as compared with 3 and 6 months)
  6. Change in the level of Protein/creatinine ratio (baseline as compared with 3 and 6 months)
  The Change in the level of Protein/creatinine ratio (baseline as compared with 3 and 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Markell, MD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No